CLINICAL TRIAL: NCT05242029
Title: A Randomized, Double-Blind Study of Psilocybin for Opioid Use Disorder in Patients on Methadone Maintenance With Ongoing Opioid Use
Brief Title: Psilocybin for Opioid Use Disorder in Patients on Methadone Maintenance With Ongoing Opioid Use
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00251861
Record Dates: First submitted 2022-02-07; First posted 2022-02-16 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to an active group or control group (46 per group). Participants will undergo a total of 2 dosing sessions (whether psilocybin or placebo). The active group will receive 40mg psilocybin first. All participants will receive a second dosing session at three months. The active group will be further randomized, with half receiving 40mg psilocybin, and half receiving placebo at three months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, and outcomes assessors will be blinded for the duration of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin (Experimental): Participants will be administered 40mg of psilocybin in a clinical setting. Psilocybin is administered orally as a capsule and taken with water.
  At 3 months, half will be randomized to receive a blinded dose of psilocybin 40mg and half a blinded dose of placebo.
  Interventions: Drug: Placebo; Drug: Psilocybin
- Placebo (Placebo Comparator): Participants will be administered placebo in a clinical setting. Placebo is administered orally as a capsule taken with water.
  At 3 months, participants will receive a blinded dose of psilocybin 40mg.
  Interventions: Drug: Placebo; Drug: Psilocybin

INTERVENTIONS:
Drug: Placebo — Participants will receive placebo in a clinical setting.
Drug: Psilocybin — Participants will receive 40mg psilocybin in a clinical setting.

SUMMARY:
This study will investigate whether psilocybin administered under supportive conditions can reduce illicit opioid use and improve quality of life in individuals with Opioid Use Disorder (OUD) in Methadone Maintenance Treatment (MMT) who are concurrently using other opioids illicitly.

DETAILED DESCRIPTION:
This randomized double-blind placebo-controlled trial will investigate whether 2 doses of psilocybin administered under supportive conditions can reduce illicit opioid use (assessed by self-report and urine toxicology) and improve quality of life as measured by World Health Organization Quality of Life (WHOQOL-BREF) in individuals with OUD in MMT who are concurrently using other opioids illicitly. In addition, the investigators will investigate secondary outcomes including whether psilocybin under supportive conditions improves mood, reduces use of tobacco and other non-opioid drugs, improves chronic pain and sleep.

Ninety-two participants aged 21-70 who meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for OUD, are enrolled in a MMT program for at least 3 months, and have urine toxicology positive for methadone and another opioid will be recruited from the community and complete all study procedures. Participants will be randomized to an active group or control group (46 per group). Participants will undergo a total of 2 dosing sessions (whether psilocybin or placebo). The active group will receive 40mg psilocybin first. All participants will receive a second dosing session at three months. The active group will be further randomized, with half receiving 40mg psilocybin, and half receiving placebo at three months to test a secondary hypothesis that two doses of psilocybin are more effective in treating OUD than a single dose.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-70 years
* Have OUD
* Enrolled in a methadone maintenance program for at least 3 months
* Urine toxicology positive for methadone
* Urine toxicology positive for an additional opioid
* Access to stable housing
* Read, write, and speak English
* Be judged by study team clinicians to be at low risk for suicidality
* Have limited lifetime use of classic psychedelics (no use in the past 5 years; total classic psychedelic use less than 20 times)
* Are local to the Baltimore area

Exclusion Criteria:

* Women who are pregnant, nursing, or not practicing an effective means of birth control
* Cardiovascular conditions: hypertension with resting blood pressure systolic >140 or diastolic >90, angina, a clinically significant ECG abnormality (e.g., atrial fibrillation, corrected QT interval > 450), transient ischemic attack in the last 6 months stroke, peripheral or pulmonary vascular disease
* Epilepsy
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking a prescribed psychoactive medication on a daily basis (except methadone)
* Currently taking on a daily basis any medications (including herbal substances and supplements) with a central nervous system effect on serotonin, including serotonin-reuptake inhibitors and monoamine oxidase inhibitors.

  o For individuals who have intermittent or as needed use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
* Currently taking efavirenz, Acetaldehyde dehydrogenase inhibitors such as disulfiram (Antabuse), Alcohol dehydrogenase inhibitors, or Uridine 5'-diphospho-glucuronosyltransferase Family 1 Member A9 (UGT1A9) inhibitors or UGT1A10 inhibitors such as phenytoin, regorafenib, eltrombopag.
* Have a seizure disorder, multiple sclerosis, history of significant head trauma, central nervous system tumor, movement disorders or any neurodegenerative condition.
* Morbidly obese (>100 lbs above idea body weight, or BMI >=40, or BMI >=35 with high blood pressure or diabetes)
* Body weight < 45kg
* Recent (within past 12 months) or extensive history of classic psychedelic use (>19 lifetime uses).
* Physiological dependence on benzodiazepines or alcohol
* Abnormal screening labs: values for hemoglobin, white blood count, creatinine, potassium, and bilirubin outside of the normal lab reference rage. Transaminases greater than x2 the upper limit of normal lab reference range.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in non-methadone opioid use as assessed by urine toxicology | Baseline and 3-months after first experimental drug administration session
  The primary outcome variable will be change in non-methadone opioid use as verified by urine toxicology at each visit.
Change in non-methadone opioid use as assessed by the Timeline Follow Back self report | Baseline and 3-months after first experimental drug administration session
  The primary outcome variable will be change in non-methadone opioid use as verified by Timeline Follow Back (TLFB) of mean number of days of non-methadone opioid use. The TLFB is a widely used, standardized, calendar-based retrospective self-report assessment to quantify daily opioid use.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Johnson, PhD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicholas CR, Horton DM, Malicki J, Baltes A, Hutson PR, Brown RT. Psilocybin for Opioid Use Disorder in Two Adults Stabilized on Buprenorphine: A Technical Report on Study Modifications and Preliminary Findings. Psychedelic Med (New Rochelle). 2023 Dec 13;1(4):253-261. doi: 10.1089/psymed.2023.0012. eCollection 2023 Dec. PMID 40046866